CLINICAL TRIAL: NCT07384702
Title: Phase 2 Platform Randomized, Multicentre and Open Trial on the Efficacy and Safety of Clopidogrel as Adjuvant Drug in Staphylococcus Aureus Bacteraemia (CLOPI-SNAP)
Brief Title: Adjuvant Clopidogrel in Staphylococcus Aureus Bacteremia
Acronym: CLOPI-SNAP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOPI-SNAP; 2023-503582-35-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bacteremia Due to Staphylococcus Aureus
Keywords: bacteriemia; Staphylococcus aureus; adjunctive treatment; Platform trial; Clopidogrel; Desirability of Outcome Ranking
MeSH Terms: conditions — Staphylococcal Infections | interventions — Clopidogrel

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized 1:1 to receive either oral clopidogrel for 5 days-administered as a 300 mg loading dose on Day 1 followed by 75 mg once daily on subsequent days-or no antiplatelet therapy (antibiotic treatment according to SNAP assignment).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral clopidogrel (Experimental): Oral clopidogrel 75 mg pills; 300 mg from domain reveal (day 1 of treatment), followed by 75 mg daily until day 5 of treatment inclusive (4 additional calendar days) added to different concurrent antibiotic options currently approved for SAB
  Interventions: Drug: Clopidogrel
- No antiplatelet treatment (Other): Patients receive different concurrent antibiotic options currently approved for SAB
  Interventions: Drug: No antiplatelet treatment

INTERVENTIONS:
Drug: Clopidogrel — Oral clopidogrel 75 mg pills; 300 mg from domain reveal (day 1 of treatment), followed by 75 mg daily until day 5 of treatment inclusive (4 additional calendar days)
  Other Names: antiplatelet arm
  Arms: Oral clopidogrel
Drug: No antiplatelet treatment — Different concurrent antibiotic options currently approved for SAB
  Arms: No antiplatelet treatment

SUMMARY:
The CLOPI-SNAP study is a randomized, multicenter, open-label clinical trial embedded within the SNAP (NCT 05137119) research platform. It constitutes a sub-study added to the core protocol for patients suffering Staphylococcus aureus bacteremia (SAB).

DETAILED DESCRIPTION:
The CLOPI-SNAP study evaluates whether the administration of clopidogrel as adjunctive therapy improves clinical outcomes while maintaining an acceptable safety profile in hospitalized patients with Staphylococcus aureus bacteremia (SAB).

To be eligible for the SNAP platform (NCT 05137119), patients must meet at least two criteria: isolation of the Staphylococcus aureus complex from ≥1 blood culture and admission to a participating hospital at the time of eligibility assessment. SNAP is designed to concurrently evaluate multiple therapeutic strategies. Patients are randomly assigned to different concurrent treatment options that are currently considered acceptable in routine clinical practice; thus, standard-of-care therapy consists of approved antibiotics for the treatment of Staphylococcus aureus infection.

Specifically, patients participating in CLOPI-SNAP-adult patients with SAB enrolled in the SNAP platform-are randomized in a 1:1 ratio to receive either oral clopidogrel for 5 days, administered as a 300-mg loading dose on Day 1 followed by 75 mg once daily on subsequent days, or no antiplatelet therapy. The primary endpoint is the Desirability of Outcome Ranking (DOOR) assessed at Day 90, a hierarchical composite outcome integrating survival, clinical failure, infectious complications, and the occurrence of serious adverse events. The limited 5-day duration of clopidogrel administration is intended to focus its potential therapeutic benefit on the early phase of infection, characterized by high bacterial burden and systemic inflammation, while minimizing the risk of bleeding associated with prolonged antiplatelet exposure.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, patients must meet the same criteria as those of the general SNAP platform, as well as the domain-specific criteria:

* Microbiological isolation: Presence of Staphylococcus aureus complex in at least one blood culture.
* Hospitalization status: The patient must be admitted to a participating hospital at the time of eligibility assessment.
* Time window: Eligibility assessment must be completed within 72 hours after collection of the initial blood culture.

Exclusion Criteria:

General Medical and Safety Factors:

* Allergies: Known hypersensitivity to thienopyridines (clopidogrel, prasugrel, ticlopidine).
* Clinical status: Inability to tolerate or take oral medications, and severe hepatic impairment (Child-Pugh Class C).
* Pregnancy: Pregnant or breastfeeding women.

High Risk of Bleeding or Hematologic Disorders:

* Active or recent bleeding: Significant bleeding or invasive procedures within the previous 7 days.
* Planned surgeries: Requirement for major surgical intervention within 10 days following study enrollment.
* Coagulation parameters: Platelet count <50,000/mm³ or known coagulation disorders.
* Concomitant medications: Patients already receiving regular aspirin therapy, other P2Y12 inhibitors, or therapeutic-dose anticoagulants (prophylactic-dose heparin is permitted).

Specific Diagnoses and Clinical Criteria:

* Endocarditis: Confirmed diagnosis or clinical suspicion of bacterial endocarditis. Sources indicate that exclusion of endocarditis is justified because the potential benefit of clopidogrel is expected during early phases of high bacterial burden, whereas bleeding risk increases with prolonged treatment or established deep-seated infections.
* Medical judgment: If the treating clinical team determines that participation in this domain is not in the patient's best interest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) | At day 90 from day 0.
  Desirability of Outcome Ranking is an ordinal scale that classifies each patient's overall clinical outcome from 1 to 5, integrating survival, clinical response, and serious adverse events. DOOR 1 represents the most favorable outcome (alive with clinical cure or improvement and no serious adverse events); DOOR 2, clinical cure or improvement with serious adverse events; DOOR 3, alive with clinical failure and no serious adverse events; DOOR 4, clinical failure with serious adverse events; and DOOR 5, death, representing the least desirable outcome. Lower numerical values indicate more favorable overall clinical outcomes.

SECONDARY OUTCOMES:
Mortality | At day 14 and day 28 from day of assignment of study drug (day 0)
  Dead of any cause
Length of stay of inpatient hospitalisation | At day 90 from day 0.
  Length of hospital stay in days from patient enrollment into the study to the time of hospital discharge or death
Microbiological treatment failure | At day 14 and day 90 from day of assignment of study drug (day 0)
  Defined as a positive S. aureus culture from a sterile site (deep tissue or abscess).
New foci of infection | At day 14 and day 90 from day of assignment of study drug (day 0)
  Diagnosis of new infection foci, based on clinical, radiological, microbiological, or pathological findings.

OTHER OUTCOMES:
Major bleeding | At day 90 from day 0.
  Defined as any bleeding that is fatal, occurs in a critical organ or area, causes a hemoglobin drop of ≥2 g/dL, or requires transfusion of ≥2 units of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodriguez Baños, PhD, Study Chair — Hospital Universitario Virgen Macarena
Locations (20):
- Spain (20):
  - Hospital General Universitario de Alicante, Alicante
  - H.U. Clinic, Barcelona
  - H.U. Mutua Terrassa, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Bellvitge, Barcelona
  - Hospital Universitario de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - H.U. Reina Sofía, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - H.U. Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario La paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Virgen Macarena, Seville
  - H.U. Virgen del Rocío, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Marqués de Valdecilla, Valdecilla
  - Hospital Universitario Álvaro Cunqueiro, Vigo
  - Hospital Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No
The information will be made available upon completion of the study. During the study period and data preparation phase, the information will be under the custody and responsibility of the research team.

REFERENCES:
- [Background] Campbell AJ, Anpalagan K, Best EJ, Britton PN, Gwee A, Hatcher J, Manley BJ, Marsh J, Webb RH, Davis JS, Mahar RK, McGlothlin A, McMullan B, Meyer M, Mora J, Murthy S, Nourse C, Papenburg J, Schwartz KL, Scheuerman O, Snelling T, Strunk T, Stark M, Voss L, Tong SYC, Bowen AC; Staphylococcus aureus Network Adaptive Platform Paediatric and Youth (SNAP-PY) working groupSNAP Global Trial Steering Committee. Whole-of-Life Inclusion in Bayesian Adaptive Platform Clinical Trials. JAMA Pediatr. 2024 Oct 1;178(10):1066-1071. doi: 10.1001/jamapediatrics.2024.2697. PMID 39158898
- [Background] Mahar RK, McGlothlin A, Dymock M, Barina L, Bonten M, Bowen A, Cheng MP, Daneman N, Goodman AL, Lee TC, Lewis RJ, Lumley T, McLean ARD, McQuilten Z, Mora J, Paterson DL, Price DJ, Roberts J, Snelling T, Tverring J, Webb SA, Yahav D, Davis JS, Tong SYC, Marsh JA; SNAP Global Trial Steering Committee. Statistical documentation for multi-disease, multi-domain platform trials: our experience with the Staphylococcus aureus Network Adaptive Platform trial. Trials. 2025 Feb 11;26(1):49. doi: 10.1186/s13063-024-08684-8. PMID 39934879
- [Background] Boyles T, Bowen AC, Chomba R, Nel J, Davis JS, Tong SYC. Inclusion of a low- and middle-income country site in the Staphylococcus aureus Network Adaptive Platform trial: experiences from Johannesburg. Clin Microbiol Infect. 2025 Dec;31(12):1948-1950. doi: 10.1016/j.cmi.2025.06.032. Epub 2025 Jul 4. No abstract available. PMID 40618922
- [Background] Walls G, McGrath L, Herdman MT, Campbell AJ, Cheng MP, Marks M, Oever JT, Sahng E, Yahav D, Tong SYC, Goodman AL, Lim AG, Bloomfield M; Staphylococcus aureus Network Adaptive Platform Trial Early Oral Switch Domain Specific Working Group. Patient-reported perceptions, experiences and preferences around intravenous and oral antibiotics for the treatment of Staphylococcus aureus bacteremia: a descriptive qualitative study. Clin Infect Dis. 2025 Sep 24:ciaf522. doi: 10.1093/cid/ciaf522. Online ahead of print. PMID 40988120
- [Background] de Kretser D, Mora J, Bloomfield M, Campbell A, Cheng MP, Guy S, Hensgens M, Kalimuddin S, Lee TC, Legg A, Mahar RK, Marks M, Marsh J, McGlothin A, Morpeth SC, Sud A, Ten Oever J, Yahav D, Bonten M, Bowen AC, Daneman N, van Hal SJ, Heriot GS, Lewis RJ, Lye DC, McQuilten Z, Paterson DL, Owen Robinson J, Roberts JA, Scarborough M, Webb SA, Whiteway L, Tong SYC, Davis JS, Walls G, Goodman AL; SNAP Early Oral Switch Domain-Specific Working Group and SNAP Global Trial Steering Committee; SNAP Trial Group. Early Oral Antibiotic Switch in Staphylococcus aureus Bacteraemia: The Staphylococcus aureus Network Adaptive Platform (SNAP) Trial Early Oral Switch Protocol. Clin Infect Dis. 2024 Oct 15;79(4):871-887. doi: 10.1093/cid/ciad666. PMID 37921609
- See also: complete Snap platform trial — http://www.snaptrial.com.au